CLINICAL TRIAL: NCT02320916
Title: A Randomized Controlled Trial on the Effect of Needle Gauge on the Pain and Anxiety Experienced During Arterial Puncture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2010/191/SC
Record Dates: First submitted 2014-12-10; First posted 2014-12-19 (Estimated); Last update posted 2016-08-17 (Estimated); Status verified 2016-08

CONDITIONS: Blood Gas Analysis; Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 23Gauge (Active Comparator): Arterial blood puncture will be performed using a 23Gauge needle
  Interventions: Procedure: 23Gauge
- 25Gauge (Active Comparator): Arterial blood puncture will be performed using a 25Gauge needle
  Interventions: Procedure: 25Gauge

INTERVENTIONS:
Procedure: 23Gauge — Arterial puncture will be made using a 23Gauge needle
  Arms: 23Gauge
Procedure: 25Gauge — Arterial puncture will be made using a 25Gauge needle
  Arms: 25Gauge

SUMMARY:
Arterial blood-gas (ABG) measurements are the gold standard to evaluate pulmonary gas exchange. However, arterial punctures are more painful than venous punctures and, in ICU patients, cause greater anxiety than tracheal aspiration. The only technique that has been shown to effectively reduce pain during arterial punctures is the subcutaneous injection of lidocaine. However, this technique is more time consuming and is poorly used.

Topical anesthesia is widely used during arterial punctures despite the lack of proof of efficacy.

While performing arterial punctures with small gauge needles is feasible, to the best of the investigators knowledge no studies have assessed the effect of needle gauge on arterial puncture related pain.

The aim of the present study was to compare the pain experienced during arterial punctures performed with a 25 G or 23 G needle. The secondary endpoints were the characterization of the pain and the anxiety associated with the arterial punctures.

ELIGIBILITY:
Inclusion Criteria:

* patients who had a planned assessment of arterial blood gas in our Respiratory Department

Exclusion Criteria:

* under the age of 18
* inability to provide consent
* the presence of a contraindication to arterial punctures based on the American Association of Respiratory Care Guidelines

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2013-04; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Pain experienced by the patient during arterial puncture | Less thant 60minutes after puncture
  Evaluated using a Visual Analogue Scale for pain. Graduated from 0 to 100mm

SECONDARY OUTCOMES:
Anxiety before and after puncture arterial puncture | Before puncture and less than 60minutes after puncture
  Evaluated using a Visual Analogue Scale for anxiety. Graduated from 0 to 100mm
Most painful moment of the arterial puncture | Less than 60minutes after puncture
  Evaluated by a standardised questionnaire: The most painful moment was :
  A/ At needle insertion B/ During puncture C/ After puncture D/ While the puncture was repeated
Duration of arterial puncture | 10minutes
  Time needed to perform the procedure will be evaluated using a chronometer. The number of seconds needed to collect the arterial blood gas will we recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Bouchra Lamia, MD, MPH, PhD, Principal Investigator — University Hospital, Rouen
Locations (1):
- CHU de Rouen, Rouen, France

REFERENCES:
- [Derived] Patout M, Lamia B, Lhuillier E, Molano LC, Viacroze C, Benhamou D, Muir JF, Cuvelier A. A Randomized Controlled Trial on the Effect of Needle Gauge on the Pain and Anxiety Experienced during Radial Arterial Puncture. PLoS One. 2015 Sep 25;10(9):e0139432. doi: 10.1371/journal.pone.0139432. eCollection 2015. PMID 26407017